CLINICAL TRIAL: NCT04776915
Title: Investigation of the Effect of Serum Androgen and Anti-Mullerian Hormone Levels on the Frequency of Müllerian Anomalies and Pregnancy Outcomes in Patients With Polycystic Ovarian Syndrome Undergoing Invitro Fertilization
Brief Title: Congenital Uterine Anomalies & Pregnancy in Polycystic Ovarian Syndrome
Acronym: CONUTA&PPCOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, GÜRKAN UNCU,PROF. MD, Prof. Dr., Uludag University
Other Study IDs: 2020-18/17
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Mullerian Anomaly of Uterus, Nec
Keywords: mullerian anomaly, PCOS, antimullerian hormone
MeSH Terms: conditions — Enterocolitis, Necrotizing; Polycystic Ovary Syndrome | interventions — Ultrasonography; Hysterosalpingography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Infertile patients due to polycystic ovarian syndrome
  Interventions: Diagnostic Test: Ultrasound and Hysterosalpingography
- Control Group: Infertile patients due to unexplained infertility
  Interventions: Diagnostic Test: Ultrasound and Hysterosalpingography

INTERVENTIONS:
Diagnostic Test: Ultrasound and Hysterosalpingography — Ultrasound and Hysterosalpingography

SUMMARY:
Prospective research in which patients who applied to UUTF Gynecology and Obstetrics ART center for the treatment of infertility (inability to conceive despite one year of unprotected sexual intercourse), who will undergo IVF due to PCOS and unexplained infertility

DETAILED DESCRIPTION:
As of 01/10/2020, IVF cycles of patients with PCOS (n = 105) and unexplained infertility (n = 105) who have applied to Bursa Uludag University Gynecology and Obstetrics Department, Reproductive Treatments Center, will be included in the study. Demographic data of all patients (age, BMI, smoking), presence of hyperandrogenism findings such as systemic diseases, hirsutism, alopecia, FSH, LH, LH/FSH ratio, estradiol levels, pregestational serum AMH levels, uterine anomalies detected by transvaginal USG or hysterosalpingography, controlled ovarian hyperstimulation protocols and doses; Besides, DHEA-S, Free Testosterone, 17-OH Progesterone levels will be recorded in patients diagnosed with PCOS. All these data are routine laboratory and imaging parameters of patients who underwent in vitro fertilization in our UYTE center. Pregnancy results of the patients (biochemical pregnancy, anembryonic pregnancy, abortion, clinical pregnancy, live birth), perinatal results and complications during clinical pregnancy, delivery ways, and newborn APGAR scores will be recorded. Results will be compared with patients in the control group diagnosed with unexplained infertility.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 20-40
* Need for an assisted reproductive method due to PCOS or unexplained infertility

Exclusion Criteria:

* <20 years or >40 years
* Detecting a cause for infertility other than PCOS

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile Patients who undergo IVF&ICSI treatment
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
The rate of Mullerian Abnormality | One year
  ESHRE&ESGE uterine abnormality classification

CONTACTS AND LOCATIONS:
Overall Officials: Özge Albayrak, M.D, Principal Investigator — Bursa Uludag University School of Medicine ART Center
Locations (1):
- Uludag University ART Center, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No